CLINICAL TRIAL: NCT05876078
Title: DORAYA-HF EU: Assessment of the Doraya Catheter for the Treatment of Volume Overload in Acute Heart Failure Patients With Insufficient Response to Diuretics
Brief Title: DORAYA-HF OUS Assessment of the Doraya Catheter for the Treatment of ADHF Patients With Insufficient Response to Diuretics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Revamp Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIS-D-04
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Decompensated Heart Failure
Keywords: ADHF

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ADHF patients (Experimental): ADHF patients with insufficient response to diuretics treated with the Doraya catheter
  Interventions: Device: Doraya catheter

INTERVENTIONS:
Device: Doraya catheter — Temporary deployment of the Doraya catheter in ADHF patients

SUMMARY:
The study objective is to evaluate the feasibility of the Doraya Catheter and measure clinical performance and safety endpoints, in ADHF patients deemed to have insufficient diuretic response.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is hospitalized with primary diagnosis of ADHF.
2. N-terminal-pro-brain natriuretic peptide (NT-proBNP) ≥1,000 pg/m orvBNP≥250 pg/mL.
3. Evidence of fluid overload.
4. Subject insufficiently responds to IV diuretic therapy

Exclusion Criteria:

Systolic blood pressure < 80 mmHg at the time of screening. 2. Acute myocardial infarction or acute coronary syndrome or cardiogenic shock or pleurocentesis within past 14 days or cardiovascular intervention within past 14 days. 3. Complex congenital heart disease (e.g., Tetralogy of Fallot subjects, single ventricle physiology).

4. Known active myocarditis, hypertrophic obstructive cardiomyopathy, infiltrative cardiomyopathy (e.g., amyloidosis), constrictive pericarditis or cardiac tamponade.

5. Severe Aortic valvular disorder (i.e., hemodynamically relevant valvular diseases such as severe stenosis \severe regurgitation) or Severe mitral disease with planned intervention.

6. Evidence of active systemic infection documented by either one of the following: fever >38°C/100°F, or ongoing uncontrolled infection (i.e., inflammatory parameters not decreasing despite > 48 hours of antibiotic treatment).

7. Moribund subject or subject with severe or deteriorating damage in more than 3 critical body systems, based on investigator's clinical judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 30 day post Doraya procedure
  Device or procedure related SAEs rate (including MACE) based on MM adjudication.
Urine Output | 24 hours pre Doraya deployment, during Doraya indwelling period, and for 24 hours after Doraya removal
  Change in total urine output

CONTACTS AND LOCATIONS:
Locations (21):
- Czechia (3):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice u sv. Anny v Brne, Brno
  - Fakultní nemocnice Hradec Králové, Hradec Králové
- Georgia (2):
  - LLC Bokhua Memorial Cardiovascular Center, Tbilisi
  - LTD Israel Georgian Medical Research Clinic Helsicore, Tbilisi
- Germany (5):
  - Herzzentrum der Universität zu Köln, Cologne
  - Heartcenter Dresden, Dresden
  - Klinikum Fürth, Fürth
  - UKSH Universitäres Herzzentrum Lübeck, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Hungary (2):
  - Semmelweis University Heart and Vascular Center, Budapest
  - University Hospital of Szeged, Szeged
- A.O.U Pisana Cisanello, Pisa, Italy
- Poland (2):
  - Narodowy Instytut Kardiologii Stefana kardynała Wyszyńskiego Państwowy Instytut Badawczy, Warsaw
  - Mikulicz-Radecki University Teaching Hospital in Wrocław, Wroclaw
- Slovakia (2):
  - SUSCCH, Banská Bystrica
  - CINRE, s.r.o., Bratislava
- Spain (4):
  - Hospital clinic de Barcelona, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided